CLINICAL TRIAL: NCT00860106
Title: Study of Predictive Echo Doppler Score and D-dimer Level in Evaluation of the Thromboembolic Event Recurrence After Anticoagulant Treatment Cessation.
Brief Title: Echo Doppler (ED )Score and D-dimer (DD) Level in the Evaluation of VTE Recurrence After Anticoagulant Treatment Cessation
Acronym: VAPRED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DCIC 04 22
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Previous Vka Treatment; Previous Proximal VTE
Keywords: VTE; VKA treatment; VKA treatment cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Follow up (Other): ED score and DDimer level of patients who have stopped their VKA treatment (after the first or the second previous proximal VTE).
  Phone follow up for 2 years.
  Interventions: Other: ED, DDimers and phone follow up

INTERVENTIONS:
Other: ED, DDimers and phone follow up — ED score, DDimers level and phone questionnary

SUMMARY:
The purpose of this trial is to perform a prospective multicentric study to determine predictive ED score and D-dimer level in the evaluation of the thromboembolic event recurrence after anticoagulant treatment cessation.

The patients are included in the study from the anticoagulant treatment cessation. An ED score and a blood sample are performed at this time and one month later. Then, the patients are followed up by phone for 2 years.

DETAILED DESCRIPTION:
DDimer levels are centralized in University Hospital of Grenoble at the end of the study

ELIGIBILITY:
Inclusion Criteria:

* > 18 and <80 years old
* First or second treated proximal VTE event (+/- Pulmonary embolism)
* Signed informed consent

Exclusion Criteria:

* Active cancer or currently treated
* Previous VTE>2
* Long term anticoagulant treatment for VTE diseases
* Long term anticoagulant treatment for other diseases
* Pregnancy, parturient or breast feeding
* Person deprived of freedom by judicial or administrative decision
* Consent unsigned

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2005-03; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
VTE event recurrence | 0-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilles PERNOD, Professor, Principal Investigator — University Hospital, Grenoble
Locations (16):
- France (16):
  - University Hospital, Amiens
  - Cabinet Medical, Annecy
  - HOSPITAL, Annecy
  - Cabinet Medical, Bourgoin
  - Cabinet Medical, Chalon-sur-Saône
  - HOSPITAL, Chambéry
  - Cabinet Medical, Crolles
  - Cabinet Medical, Fontaine
  - Vascular Medecine Departement - University Hospital of Grenoble, Grenoble
  - Cabinet Medical, Grenoble
  - Clinique Mutualiste les eaux claires, Grenoble
  - Cabinet Medical, Meylan
  - Cabinet Medical, Pontcharra
  - Cabinet Medical, Saint-Égrève
  - CMC Les Petites Roches, Saint-Hilaire
  - Cabinet Medical, Voiron

REFERENCES:
- [Background] Agnelli G, Prandoni P, Santamaria MG, Bagatella P, Iorio A, Bazzan M, Moia M, Guazzaloca G, Bertoldi A, Tomasi C, Scannapieco G, Ageno W; Warfarin Optimal Duration Italian Trial Investigators. Three months versus one year of oral anticoagulant therapy for idiopathic deep venous thrombosis. Warfarin Optimal Duration Italian Trial Investigators. N Engl J Med. 2001 Jul 19;345(3):165-9. doi: 10.1056/NEJM200107193450302. PMID 11463010
- [Background] Agnelli G, Prandoni P, Becattini C, Silingardi M, Taliani MR, Miccio M, Imberti D, Poggio R, Ageno W, Pogliani E, Porro F, Zonzin P; Warfarin Optimal Duration Italian Trial Investigators. Extended oral anticoagulant therapy after a first episode of pulmonary embolism. Ann Intern Med. 2003 Jul 1;139(1):19-25. doi: 10.7326/0003-4819-139-1-200307010-00008. PMID 12834314
- [Background] Bosson JL, Riachi M, Pichot O, Michoud E, Carpentier PH, Franco A. Diameters of acute proximal and distal deep venous thrombosis of the lower limbs. Int Angiol. 1998 Dec;17(4):260-7. PMID 10204659
- [Background] Cushman M, Folsom AR, Wang L, Aleksic N, Rosamond WD, Tracy RP, Heckbert SR. Fibrin fragment D-dimer and the risk of future venous thrombosis. Blood. 2003 Feb 15;101(4):1243-8. doi: 10.1182/blood-2002-05-1416. Epub 2002 Sep 26. PMID 12393393
- [Background] Eichinger S, Minar E, Bialonczyk C, Hirschl M, Quehenberger P, Schneider B, Weltermann A, Wagner O, Kyrle PA. D-dimer levels and risk of recurrent venous thromboembolism. JAMA. 2003 Aug 27;290(8):1071-4. doi: 10.1001/jama.290.8.1071. PMID 12941680
- [Background] Emmerich J, Fiessinger JN. Residual venous thrombosis and recurrent thromboembolism. Ann Intern Med. 2003 Aug 19;139(4):303; author reply 304. doi: 10.7326/0003-4819-139-4-200308190-00017. No abstract available. PMID 12965991
- [Background] Fattorini A, Crippa L, Vigano' D'Angelo S, Pattarini E, D'Angelo A. Risk of deep vein thrombosis recurrence: high negative predictive value of D-dimer performed during oral anticoagulation. Thromb Haemost. 2002 Jul;88(1):162-3. No abstract available. PMID 12152661
- [Background] Kearon C, Gent M, Hirsh J, Weitz J, Kovacs MJ, Anderson DR, Turpie AG, Green D, Ginsberg JS, Wells P, MacKinnon B, Julian JA. A comparison of three months of anticoagulation with extended anticoagulation for a first episode of idiopathic venous thromboembolism. N Engl J Med. 1999 Mar 25;340(12):901-7. doi: 10.1056/NEJM199903253401201. PMID 10089183
- [Background] Kuruvilla J, Wells PS, Morrow B, MacKinnon K, Keeney M, Kovacs MJ. Prospective assessment of the natural history of positive D-dimer results in persons with acute venous thromboembolism (DVT or PE). Thromb Haemost. 2003 Feb;89(2):284-7. PMID 12574808
- [Background] Palareti G, Legnani C, Cosmi B, Guazzaloca G, Pancani C, Coccheri S. Risk of venous thromboembolism recurrence: high negative predictive value of D-dimer performed after oral anticoagulation is stopped. Thromb Haemost. 2002 Jan;87(1):7-12. PMID 11848459
- [Background] Palareti G, Legnani C, Cosmi B, Valdre L, Lunghi B, Bernardi F, Coccheri S. Predictive value of D-dimer test for recurrent venous thromboembolism after anticoagulation withdrawal in subjects with a previous idiopathic event and in carriers of congenital thrombophilia. Circulation. 2003 Jul 22;108(3):313-8. doi: 10.1161/01.CIR.0000079162.69615.0F. Epub 2003 Jul 7. PMID 12847064
- [Background] Pernod G, Mossuz P, Polack B. Optimized factor V gene mutation detection using buffy-coat direct PCR. Biotechniques. 1997 May;22(5):837, 840, 841. doi: 10.2144/97225bm10. No abstract available. PMID 9149858
- [Background] Piovella F, Crippa L, Barone M, Vigano D'Angelo S, Serafini S, Galli L, Beltrametti C, D'Angelo A. Normalization rates of compression ultrasonography in patients with a first episode of deep vein thrombosis of the lower limbs: association with recurrence and new thrombosis. Haematologica. 2002 May;87(5):515-22. PMID 12010666
- [Background] Prandoni P, Lensing AW, Prins MH, Bernardi E, Marchiori A, Bagatella P, Frulla M, Mosena L, Tormene D, Piccioli A, Simioni P, Girolami A. Residual venous thrombosis as a predictive factor of recurrent venous thromboembolism. Ann Intern Med. 2002 Dec 17;137(12):955-60. doi: 10.7326/0003-4819-137-12-200212170-00008. PMID 12484710
- [Background] Schulman S, Rhedin AS, Lindmarker P, Carlsson A, Larfars G, Nicol P, Loogna E, Svensson E, Ljungberg B, Walter H. A comparison of six weeks with six months of oral anticoagulant therapy after a first episode of venous thromboembolism. Duration of Anticoagulation Trial Study Group. N Engl J Med. 1995 Jun 22;332(25):1661-5. doi: 10.1056/NEJM199506223322501. PMID 7760866
- [Background] Schulman S, Granqvist S, Holmstrom M, Carlsson A, Lindmarker P, Nicol P, Eklund SG, Nordlander S, Larfars G, Leijd B, Linder O, Loogna E. The duration of oral anticoagulant therapy after a second episode of venous thromboembolism. The Duration of Anticoagulation Trial Study Group. N Engl J Med. 1997 Feb 6;336(6):393-8. doi: 10.1056/NEJM199702063360601. PMID 9010144
- [Background] Schulman S. Clinical practice. Care of patients receiving long-term anticoagulant therapy. N Engl J Med. 2003 Aug 14;349(7):675-83. doi: 10.1056/NEJMcp025373. No abstract available. PMID 12917305
- [Background] Sebastian JL, Torre DM. Residual venous thrombosis and recurrent thromboembolism. Ann Intern Med. 2003 Aug 19;139(4):303; author reply 304. doi: 10.7326/0003-4819-139-4-200308190-00016. No abstract available. PMID 12965989